CLINICAL TRIAL: NCT06805214
Title: Increased Body Temperature Post Tracheostomy: a Retrospective Study
Status: Recruiting | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, sara dichtwald, Dr, Meir Medical Center
Other Study IDs: 0021-25-MMC
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Tracheostomy Complication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: post tracheostomy fever — incidence of post tracheostomy fever and whether retrospectively the increased temperature indicated development of sepsis or not (no intervention)

SUMMARY:
Tracheostomy is one of the most common procedures in intensive care units. Post-tracheostomy increased body temperature within 24 hours is common. However, frequently sepsis workup is performed along with initiation of broad spectrum antibiotic therapy. We will investigate the incidence of post tracheostomy fever and whether retrospectively the increased temperature indicated development of sepsis or not. The study is retrospective and will be based on data collection.

ELIGIBILITY:
Inclusion Criteria: Patients admitted to the ICU from 1.2020 to 1.2025 who underwent tracheostomy during ICU admission -

Exclusion Criteria: Patients who did not fullfil the above criteria

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU from 1.2020 to 1.2025 who underwent tracheostomy during ICU admission
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Post tracheostomy fever | 24 hours post tracheostomy
  Incidence of post tracheostomy fever

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No